CLINICAL TRIAL: NCT00596895
Title: Phase II Trial of Isoflavone in Prostate-specific Antigen Recurrent Prostate Cancer After Previous Local Therapy.
Brief Title: Isoflavone in Prostate-specific Antigen Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFJ2003-113
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2008-01

CONDITIONS: Biochemical Recurrent Prostate Cancer
Keywords: Isoflavone, PSA, prostate cancer, recurrent, quality of life
MeSH Terms: conditions — Salivary Gland Adenoma, Pleomorphic; Prostatic Neoplasms; Recurrence | interventions — Isoflavones; Soy Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Isoflavone treatment
  Interventions: Dietary Supplement: Isoflavone

INTERVENTIONS:
Dietary Supplement: Isoflavone — Ingested 47 mg of isoflavone in three 8 oz servings per day
  Other Names: Soy Dream Enriched, Original or Vanilla, soy milk

SUMMARY:
Primary Outcome Measures:

Decrease in rate of serum PSA rise

Secondary Outcome Measures:

Adherence to treatment regimens

Quality of life as assessed by FACT-P at baseline and at 12 months of treatment

Modulation of serum testosterone,isoflavone metabolites, and cholesterol

Estimated Enrollment: 27 Study Start Date: November 2003 Estimated Primary Completion Date: February 2007 (Final data collection date for primary outcome measure)

DETAILED DESCRIPTION:
* Pretreatment evaluation included a complete medical history, physical examination (including digital rectal examination), serum PSA, free/total testosterone, lipids, serum isoflavone levels (genistein, daidzein, and equol), and assessment of quality of life (Functional Assessment of Cancer Treatment-Prostate, FACT-P questionnaire).
* Whole blood will be obtained prior to initiation of the study to assess for DNA polymorphism.
* Follow-up serum PSA levels to assess efficacy were obtained at 3, 6, 9, and 12 months after initiation of treatment.
* Medical history, physical examination, serum testosterone, lipids, isoflavone, and quality of life were assessed at 6 and 12 months after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Raising serum PSA profile after previous definitive therapy (e.g., radical prostatectomy or external beam radiation therapy).
* Life expectancy of at least one year and performance status of <2 of Zubrod scale.

Exclusion Criteria:

* Metastatic or locally recurrent disease demonstrated on bone scan, computed tomography or transrectal ultrasound, or be clinically symptomatic at the time of enrollment
* No androgen deprivation therapy (ADT) or chemotherapy within 12 months of entry into the study.
* Known allergic reaction to milk or soy products were excluded.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Assess the effect of soy protein/isoflavones serum PSA levels in patients previously treated with radical prostatectomy and external beam radiation therapy. | Baseline, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Assess the effect of soy protein/isoflavones on serum testosterone, isoflavone metabolites, and cholesterol. Assess the effect of soy protein/isoflavones on quality of life of these patients. | Baseline, 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles J. Rosser, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Shands, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Pendleton JM, Tan WW, Anai S, Chang M, Hou W, Shiverick KT, Rosser CJ. Phase II trial of isoflavone in prostate-specific antigen recurrent prostate cancer after previous local therapy. BMC Cancer. 2008 May 11;8:132. doi: 10.1186/1471-2407-8-132. PMID 18471323